CLINICAL TRIAL: NCT06543927
Title: Frequncy and Risk Factors of Bleeding in Patients With Chronic Kidney Disease Receiving Antigoagulants
Brief Title: Frequency and Risk Factors of Bleeding in Patients With Chronic Kidney Disease Receiving Anticoagulants
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Abozaid, Resident-internal medecine department-sohag hospital university, Sohag University
Other Study IDs: Soh-Med-24-07-02MS
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases Receiving Anticoagulants
MeSH Terms: interventions — International Normalized Ratio

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: hemodialysis dependant
  Interventions: Diagnostic Test: serum creatinine; Diagnostic Test: INR
- group B: hemodialysis non dependant
  Interventions: Diagnostic Test: serum creatinine; Diagnostic Test: INR

INTERVENTIONS:
Diagnostic Test: serum creatinine — Detection of renal impairment in patients receiving anticoagulants
Diagnostic Test: INR — Detection of bleeding in patients with choronic kidney disease receiving anticoagulants

SUMMARY:
1-Introduction: Chronic kidney disease (CKD) is a significant global public health issue, closely linked to cardiovascular disease (CVD). Moreover, CKD is acknowledged as an independent risk factor for developing CVD and represents a heigh risk factor to thromboembolic disease in coronary and cerebral arteries also in the venous circulation that requires anticoagulation (1). According to the latest United States Renal Data System report, the prevalence of any CVD in CKD patients is nearly double that of the general population, at 69.8% compared to 34.8% (2). Also, if microalbuminuria is detected and glomerular filtration rate (eGFR) is less than <60 mL/min/1.73m2, there is an increased risk of cardiovascular events, venous thrombosis and mortality (3).

On the other hand, patients with an eGFR of less than 60 mL/min/1.73m² have double the risk of atrial fibrillation (AF) and acute coronary syndrome (ACS) (4&5). For dialysis-dependent CKD patients, the prevalence of AF is 11.6%, and within 12 months after kidney transplantation, the risk of AF occurrence rises to 35.6% per 1000 patient-years (6). Also, the risk of pulmonary venous thromboembolism (VTE) in CKD increases by 25%-30% is constant in all CKD stages, and typically characterizes the nephrotic syndrome (7).

Oral anticoagulant is an effective mean of reducing rate of ischemic stroke and systemic embolism in patient with AF in CKD patient and minimizing the morbidity and the mortality caused by venous thromboembolic disease (1). At the same time abnormalities in the platelet membrane and impaired platelet-vessel wall interaction put CKD patients at risk of bleeding significantly more than other patients of chronic disease (8).

The paradox in CKD is the association between the high thromboembolic risk and major hemorrhagic risk with declining kidney function. In CKD, managing the delicate balance between preventing thromboembolic events and avoiding hemorrhage poses significant challenges for anticoagulation treatment. This difficulty arises due to several factors:

* A higher need for anticoagulants in CKD patients.
* The absence of reliable risk scores for thromboembolic and hemorrhagic events specific to CKD patients.
* The risk-benefit ratio being influenced by numerous variables unique to this subgroup.
* Drugs bioavailability and pharmacokinetics are altered in this setting.
* A lack of consensus on recommendations for oral anticoagulation, particularly for patients in stages 4 and 5 of CKD (1).
* Randomized trials comparing direct oral anticoagulants (DOACs) and warfarin have excluded patients with creatinine clearance (CrCl) below 30 mL/min. Lack of high-quality evidence in CKD has led to differences in recommendations by various professional bodies adding on to this confusion (9). This has thus led to underutilization of DOACs in CKD patients (10) .

Due to the currently limited data, clinicians need practical clues for monitoring and optimizing the anticoagulant therapy. We try to explain the complex thrombotic-hemorrhagic state of CKD patients, and practical considerations for the management of anticoagulation in them with a focus on risk factors for bleeding.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with CKD who required and are currently receiving anticoagulation therapy according to the last guidelines, like: Patient was diagnosed with acute DVT, and or pulmonary embolism, and or splanchnic venous thrombosis.

Mechanical heart valve,

Prevention of stroke and systemic embolism in nonvalvular AF with at least one stroke risk factor :

* Prior stroke (ischaemic or unknown type), transient ischaemic attack (TIA) or non-central nervous system (CNS) systemic embolism.
* Age ≥ 75 years.
* Hypertension. iv. Diabetes mellitus.
* Heart failure and/ or left ventricular EF ≤ 35%.

  * Patients with CKD ( maintenance or not on hemodialysis)
  * Willing and agreed to be included in the study

Exclusion Criteria:

* • Significant inherited or acquired bleeding disorder

  * Patient with family history of bleeding tendency
  * Patient with contraindication to use anticoagulants
* Clinically significant active bleeding
* Hepatic disease with associated coagulopathy including Child-Pugh C
* Lesions or conditions at significant risk of bleeding including intracranial hemorrhage unless under the advice of a neurologist/neurosurgeon

  * Pregnancy, and lactating patient or suspected of pregnancy,
  * Incapable of consenting

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: • Patients with CKD who required and are currently receiving anticoagulation therapy according to the last guidelines, like: Patient was diagnosed with acute DVT, and or pulmonary embolism, and or splanchnic venous thrombosis.
  Mechanical heart valve,
  Prevention of stroke and systemic embolism in nonvalvular AF with at least one stroke risk factor :
  * Prior stroke (ischaemic or unknown type), transient ischaemic attack (TIA) or non-central nervous system (CNS) systemic embolism.
  * Age ≥ 75 years.
  * Hypertension. iv. Diabetes mellitus.
  * Heart failure and/ or left ventricular EF ≤ 35%.
    * Patients with CKD ( maintenance or not on hemodialysis)
    * Willing and agreed to be included in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
frequency of bleeding in patients with choronic kidney disease receiving anticoagulants | 6 months
  frequency and risk factors of bleeding in patients with choronic kidney disease receiving anticoagulants

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Hughes S, Szeki I, Nash MJ, Thachil J. Anticoagulation in chronic kidney disease patients-the practical aspects. Clin Kidney J. 2014 Oct;7(5):442-9. doi: 10.1093/ckj/sfu080. Epub 2014 Aug 2. PMID 25878775
- [Background] Said S, Hernandez GT. The link between chronic kidney disease and cardiovascular disease. J Nephropathol. 2014 Jul;3(3):99-104. doi: 10.12860/jnp.2014.19. Epub 2014 Jul 1. PMID 25093157
- [Background] Lau YC, Proietti M, Guiducci E, Blann AD, Lip GYH. Atrial Fibrillation and Thromboembolism in Patients With Chronic Kidney Disease. J Am Coll Cardiol. 2016 Sep 27;68(13):1452-1464. doi: 10.1016/j.jacc.2016.06.057. PMID 27659468
- [Background] Liao JN, Chao TF, Liu CJ, Wang KL, Chen SJ, Lin YJ, Chang SL, Lo LW, Hu YF, Tuan TC, Chung FP, Chen TJ, Chen SA. Incidence and risk factors for new-onset atrial fibrillation among patients with end-stage renal disease undergoing renal replacement therapy. Kidney Int. 2015 Jun;87(6):1209-15. doi: 10.1038/ki.2014.393. Epub 2015 Jan 14. PMID 25587708